CLINICAL TRIAL: NCT07299630
Title: Efficacy of Intranasal Sphenopalatine Ganglion Block by Lidocaine Spray for Partial Turbinectomy Surgeries
Brief Title: Blocking Sphenopalatine Ganglion by Intranasal Lidocaine Spray in Partial Turbinectomy Surgeries
Acronym: SPG block
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R239/2025
Record Dates: First submitted 2025-12-03; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Turbinate Surgery; Sphenopalatine Block
Keywords: SPG block; lidocaine spray; partial turbinectomy surgery
MeSH Terms: interventions — Balanced Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balanced anaesthesia (Active Comparator): Analgesia will be offered by fentanyl in induction according to Actual Body Weight (ABW). and morphine after intubation
  Interventions: Drug: Balanced anesthesia
- Lidocaine spray (Experimental): o Analgesia will be offered by fentanyl in induction according to Actual Body Weight (ABW) and then Lignocaine spray 10% 10 puffs will be applied on to the nasal cavity after directing the spray applicator parallel to the nasal floor until resistance is felt after intubation and application of nasal decongestant, in the two nostrils
  Interventions: Drug: Lidocaine spray

INTERVENTIONS:
Drug: Balanced anesthesia — Analgesia will be offered by fentanyl in induction according to Actual Body Weight (ABW). and morphine after intubation
  Arms: balanced anaesthesia
Drug: Lidocaine spray — o Analgesia will be offered by fentanyl in induction according to Actual Body Weight (ABW) and then Lignocaine spray 10% 10 puffs will be applied on to the nasal cavity after directing the spray applicator parallel to the nasal floor until resistance is felt after intubation and application of nasal decongestant, in the two nostrils
  Arms: Lidocaine spray

SUMMARY:
Nasal turbinectomy surgeries are usually done as day case surgeries as most patients are young with unremarkable comorbidities. However, considerations are still present towards patients of old age or those suffering from obesity or obstructive sleep apnea (OSA). Different techniques are still evolving to improve handling those patients to decrease complications, enhance recovery after surgery and increase patient satisfaction. Targeting sphenopalatine ganglion block by topical local anesthesia is a proposed technique that could help by decreasing peri-operative opioid consumption.

DETAILED DESCRIPTION:
Patients undergoing turbinectomy usually suffer from chronic nasal congestion with wide spectrum of symptoms ranging from headache and breathing difficulty to sleep disorders and obstructive sleep apnea that could affect daily life .

Usually the surgery is done as a day case surgery in patients without major comorbidities. Points of concern to achieve smooth outcome and enhance recovery include pain management, better surgical field for both patient and surgeon satisfaction. One approach for these goals include regional nerve blocks for the innervation of the nose .

Spheno Palatine Ganglion (SPG) block was tested with a good results for blocking autonomic innervation and subsequent decrease in pain and opioid consumption. Blockage of SPG has many approaches either trans nasal or trans oral but both are invasive and needs trained hands to do Locally infiltrating lidocaine over nasal mucosa either by lidocaine spray or a lidocaine soaked gauze was also tested in nasal surgeries with good results but doubts about duration of action of lidocaine spray is a concern that may affect post-operative pain management Targeting SPG noninvasively by lidocaine spray is proposed technique that may offer easier approach for this type of surgeries. Although concerns about effectiveness of the spray to reach and block SPG was raised before , many studies examined this approach to control headache or trigeminal neuralgia with great success.

ELIGIBILITY:
Inclusion Criteria:

• Undergoing elective partial turbinectomy surgery

Exclusion Criteria:

* Patient refusal
* Kidney or liver impairment
* Pregnant or breast-feeding women
* Allergy to any of the drugs used in the study
* OR time more than 90 min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
fentanyl doses | intraoperative
  Total doses of fentanyl rescue doses intraoperative

SECONDARY OUTCOMES:
Visual analog Score | up to 12 hours post operative
  VAS score post operative

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP